CLINICAL TRIAL: NCT07067437
Title: Single-Fraction Very Accelerated Partial Breast Irradiation (sfVAPBI) in Low-Risk Invasive or Ductal In Situ Breast Carcinoma - Phase II Multicenter Trial
Brief Title: Single-Fraction Very Accelerated Partial Breast Irradiation (sfVAPBI)
Acronym: sfVAPBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Viktor Smanykó, MD, PhD, chief physician, National Institute of Oncology, Hungary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEC-ESTRO sfVAPBI; 1012 (Registry Identifier: NNGYK)
Record Dates: First submitted 2025-06-25; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-fraction very accelerated partial breast irradiation arm (Experimental): Low risk, early-stage breast cancer patients, who receiving single-fraction very accelerated partial breast irradiation, as postoperative radiation therapy.
  Interventions: Radiation: single-fraction very accelerated partial breast irradiation

INTERVENTIONS:
Radiation: single-fraction very accelerated partial breast irradiation — Adjuvant accelerated partial breast brachytherapy, with interstitial multicatheter technique, in one fraction.

SUMMARY:
To investigate clinical outcomes, late side effects, and cosmetic results of a single-fraction very accelerated partial breast irradiation as postoperative local treatment for the treatment of early stage breast cancer.

DETAILED DESCRIPTION:
Accelerated Partial Breast Irradiation (APBI) has demonstrated the non-inferiority compared to external beam radiotherapy (EBRT) in the conserving-treatment of early breast carcinoma by using high-dose-rate (HDR) multicatheter interstitial brachytherapy (MIBT). The standard treatment regimen is 7-8 sessions with two treatments per day, for a total treatment time of 4-5 days. Based on 5-year results of the Groupe Européen de Curiethérapie European SocieTy for Radiotherapy & Oncology (GEC-ESTRO) Very Accelerated Partial Breast Irradiation (VAPBI) phase I-II trial, in low-risk cases, 3-4 fractions delivered in 2 days reduced the overall treatment time with low rate of side effects and excellent oncological outcome.

Retrospective and prospective studies with a single fraction HDR MIBT-based VAPBI suggest that by further increasing the dose delivered in one fraction, the total treatment time can be reduced to a single session safely.

A phase II multicenter trial is proposed to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0 & I & II (< 3 cm) breast carcinoma
* Lesions of < 3 cm diameter
* Invasive carcinoma of any subtype and grade or ductal carcinoma in situ (DCIS)
* Nodal status: node-negative (pN0) or micro-metastatic (pN1mi) (patients with pN1mi status can be treated, but due to the limited clinical evidence, individual decision is needed)
* M0: Absence of distant metastasis
* Clear resection margins by National Surgical Adjuvant Breast and Bowel Project (NSABP) definition (no tumor on ink)
* Unifocal (multifocality limited within 2 cm) and unicentric breast cancer
* Age> 40 years
* Luminal A or B tumors
* Time interval from surgery preferably less than 12 weeks and no longer than 20 weeks, and from adjuvant chemotherapy less than 4 weeks
* Human Epidermal growth factor Receptor 2 positive (HER2+) patients receiving postoperative anti-HER2 systemic therapy
* Specific signed consent form prior to randomization

Exclusion Criteria:

* Stage III-IV breast cancer
* Surgical margins that cannot be microscopically assessed
* Extensive intraductal component (EIC+)
* Extensive lymphovascular invasion (LVI+) (focal is allowed)
* Triple negative breast cancer
* BReast CAncer gene (BRCA) 1-2 mutation
* Human Epidermal growth factor Receptor 2 positive (HER2+) patients not receiving postoperative anti-HER2 systemic therapy
* Neoadjuvant systemic therapy
* Paget's disease or pathological skin involvement
* Synchronous or previous breast cancer.
* Pregnant or lactating women

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We can only treat female breast cancer patients with this technique.
Enrollment: 250 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Five-year incidence of late grade ≥ 2 side effects | From the third month of treatment to the end of the fifth year of follow-up.
  Radiation side effects based on Common Terminology Criteria for Adverse Events (CTCAE) (grade 1 to grade 5, higher score worse); and with the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/EORTC) Late Radiation Morbidity Scoring Schema (grade 1 to grade 4, higher score worse).

SECONDARY OUTCOMES:
Incidence (5-year actuarial rate) of ipsilateral breast recurrence (IBR) | From treatment to the end of the fifth year of follow-up.
Incidence (5-year actuarial rate) of regional relapse (RR) | From treatment to the end of the fifth year of follow-up.
Incidence (5-year actuarial rate) of contralateral breast cancer (CBC) | From treatment to the end of the fifth year of follow-up.
Incidence (5-year actuarial rate) of distant metastasis (DM) | From treatment to the end of the fifth year of follow-up.
Incidence (5-year actuarial rate) of any relapse (local, regional or distant, whichever came first) for disease free survival (DFS) | From treatment to the end of the fifth year of follow-up.
Incidence (5-year actuarial rate) of breast cancer death for cause specific survival (CSS) | From treatment to the end of the fifth year of follow-up.
Incidence (5-year actuarial rate) of death by any cause for overall survival (OS) | From treatment to the end of the fifth year of follow-up.
Incidence of acute side effects | From treatment to the end of the first 3 months of follow-up.
  Radiation side effects based on Common Terminology Criteria for Adverse Events (CTCAE) (grade 1 to grade 5, higher score worse); and with the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/EORTC) Late Radiation Morbidity Scoring Schema (grade 1 to grade 4, higher score worse).
Cosmetic results at 5 years | From treatment to the end of the fifth year of follow-up.
  Cosmetic results based on the Harvard criteria (excellent, good, fair, poor).
Quality of Life (QoL) | From treatment to the end of the fifth year of follow-up.
  European Organisation For Research And Treatment Of Cancer (EORTC) Quality of Life questionnaire (QLQ) C30 questionaire including the Breast cancer module (QLQ-BR23) (53 questions in total, from 1 to 4 points, higher score worse)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Smanykó, MD, Principal Investigator — National Institute of Oncology, Budapest, Hungary
Locations (22):
- France (3):
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Lorraine, Nancy
  - Antoine Lacassagne Cancer Centre, Nice
- Germany (5):
  - Klinikum Bremerhaven, Bremerhaven
  - University Hospital Erlangen, Erlangen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Sana Klinikum Offenbach, Offenbach
  - Universitätsklinikum Würzburg, Würzburg
- National Institute of Oncology, Budapest, Hungary
- National Cancer Institute, Vilnius, Lithuania
- Poland (5):
  - Maria Skłodowska-Curie Bialystok Oncology Center, Bialystok
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny, Brzozów
  - National Institute of Oncology, Gliwice
  - Greater Poland Cancer Centre, Poznan
  - Lower Silesian Oncology, Pulmonology and Hematology Center, Wroclaw
- Instituto Português de Oncologia do Porto, Porto, Portugal
- Oncology Institute Vojvodina, Kamenica, Serbia
- Spain (4):
  - Fundacion IMOR's Oncology Clinic, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario de Navarra, Pamplona
  - Instituto Valenciano de Oncologia, Valencia
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
3-letter abbreviation of the city of the treating hospital. Identification number of the treated patient. Performance score. Detailed histological characteristics of the breast cancer. Data of surgery and brachytherapy. Dosimetrical data. Cosmesis. Side effects. Oncological outcomes.
Supporting Information: Study Protocol
Time Frame: From treatment to the end of the 5-year follow-up period
Access Criteria: The data will be accessible to the study leader and the mathematician who prepares the statistics. The data will be transmitted encrypted to the data processing center.

REFERENCES:
- [Background] Hannoun-Levi JM, Montagne L, Sumodhee S, Schiappa R, Boulahssass R, Gautier M, Gal J, Chand ME. APBI Versus Ultra-APBI in the Elderly With Low-Risk Breast Cancer: A Comparative Analysis of Oncological Outcome and Late Toxicity. Int J Radiat Oncol Biol Phys. 2021 Sep 1;111(1):56-67. doi: 10.1016/j.ijrobp.2021.03.052. Epub 2021 Apr 6. PMID 33831490
- [Background] Hannoun-Levi JM, Gimeno Morales M, Gal J, Anchuelo J, Guinot JL, Gaztanaga M, Meszaros N, Polgar C, Strnad V, Schiappa R, Gutierrez C. Very accelerated partial breast irradiation in 1 or 2 days: Late toxicity and early oncological outcome of the GEC-ESTRO VAPBI cohort. Radiother Oncol. 2024 May;194:110217. doi: 10.1016/j.radonc.2024.110217. Epub 2024 Mar 8. PMID 38460552
- [Background] Hannoun-Levi JM, Lam Cham Kee D, Gal J, Schiappa R, Hannoun A, Fouche Y, Gautier M, Boulahssass R, Chand ME. Accelerated partial breast irradiation in the elderly: 5-Year results of the single fraction elderly breast irradiation (SiFEBI) phase I/II trial. Brachytherapy. 2020 Jan-Feb;19(1):90-96. doi: 10.1016/j.brachy.2019.10.007. Epub 2019 Nov 23. PMID 31767533
- [Background] Guinot JL, Gutierrez-Miguelez C, Meszaros N, Gonzalez-Perez V, Santos MA, Najjari D, Slocker A, Major T, Polgar C. Five-year results of the very accelerated partial breast irradiation VAPBI phase I-II GEC-ESTRO trial. Radiother Oncol. 2024 Dec;201:110543. doi: 10.1016/j.radonc.2024.110543. Epub 2024 Sep 24. PMID 39321957
- [Background] Strnad V, Polgar C, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Fietkau R, Schlamann A, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Dunst J, Gall C, Uter W; Groupe Europeen de Curietherapie and European Society for Radiotherapy and Oncology. Accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy compared with whole-breast irradiation with boost for early breast cancer: 10-year results of a GEC-ESTRO randomised, phase 3, non-inferiority trial. Lancet Oncol. 2023 Mar;24(3):262-272. doi: 10.1016/S1470-2045(23)00018-9. Epub 2023 Feb 1. PMID 36738756

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT07067437/Prot_SAP_ICF_000.pdf